CLINICAL TRIAL: NCT05654155
Title: A Pilot Study of the Feasibility and Effectiveness of Auricular Acupressure in Managing Sleep Quality, Mood Status, and Quality of Life in Parents of Children With Cancer
Brief Title: The Effectiveness of Auricular Acupressure on Sleep Quality, Mood Status, and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University of Science and Technology (Other)
Collaborators: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yi-Chien Chiang, Associate professor, Chang Gung University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMRPF1H0081
Record Dates: First submitted 2022-11-10; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Parents of Children With Cancer
Keywords: sleep quality; quality of life; auricular acupressure
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The auricular acupressure group (AAG) participants received auricular acupressure three times a day for five days every week for three weeks. Using Dr. Huang's ear reflex theory, our AAG intervention included six acupoints (i.e., shenmen, subcortex, heart, kidney, anxious, and neurasthenia points) that have been demonstrated to be effective in improving sleep and emotional stability. Participants in SAG (sham auricular acupressure group) received the same protocol of auricular acupressure as the AAG, but six acupoints were used near the treated acupoints (e.g., sacroiliac, neck, stomach, wrist, tonsil, and tongue), which would have had no effects on participants' sleep and mood status.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular acupressure group (Experimental): The AAG participants received auricular acupressure three times a day for five days every week for three weeks. Using Dr. Huang's ear reflex theory, our AAG intervention included six acupoints (i.e., shenmen, subcortex, heart, kidney, anxious, and neurasthenia points) that have been demonstrated to be effective in improving sleep and emotional stability.
  Interventions: Other: auricular acupressure
- sham auricular acupressure group (Sham Comparator): Participants in SAG received the same protocol of auricular acupressure as the AAG, but six acupoints were used near the treated acupoints (e.g., sacroiliac, neck, stomach, wrist, tonsil, and tongue), which would have had no effects on participants' sleep and mood status.
  Interventions: Other: auricular acupressure

INTERVENTIONS:
Other: auricular acupressure — Auricular acupressure therapy is a well-established treatment strategy whose foundations lie in Traditional Chinese Medicine and is a therapy that is increasingly used in Western medicine.

SUMMARY:
This pilot study aimed to determine the feasibility and effectiveness of an auricular acupressure intervention on sleep, mood state, and QOL among parents of children with cancer.

DETAILED DESCRIPTION:
This was a feasibility pilot study conducted using a randomized controlled design in which participants were randomly assigned to either an active auricular acupressure group (AAG) or a sham auricular acupressure group (SAG). Data were collected at baseline (time 0), and 1-week (time 1), 2-weeks (time 2) and 3-weeks (time 3) after the end of the intervention, which was 3 weeks long.

Participants To be included in the study, participants needed to be a parent of a child (less than 18 years old) who was newly diagnosed with cancer (less than 3 months) and who was receiving treatment with chemotherapy. Parents were excluded if they were: (1) receiving any medication or treatment for insomnia; (2) had received any acupuncture or acupressure in the recent 3 months; or (3) had ever been diagnosed with other chronic illnesses (such as cancer, heart disease, or asthma) at the time of data collection. The reason for excluding parents with chronic illnesses was to increase the similarity of subjects in this study, because such chronic illnesses may have an impact on sleep and mood.

Intervention: auricular acupressure program The AAG participants received auricular acupressure three times a day for five days every week for three weeks. Using Dr. Huang's ear reflex theory, our AAG intervention included six acupoints (i.e., shenmen, subcortex, heart, kidney, anxious, and neurasthenia points) that have been demonstrated to be effective in improving sleep and emotional stability 17, 18. Participants in SAG received the same protocol of auricular acupressure as the AAG, but six acupoints were used near the treated acupoints (e.g., sacroiliac, neck, stomach, wrist, tonsil, and tongue), which would have had no effects on participants' sleep and mood status.

Both acupressure interventions were started by cleaning the earlobe using 75% alcohol. Then, a small piece of adhesive tape with 2 seeds, which provide pressure at specific points was taped onto each selected auricular acupoint on a participant's ear. Next, the auricular therapist demonstrated the acupoints press technique to participants. The participants were asked to press one acupoint slightly to more firmly for 1 minute by themselves until they felt discomfort or tingling, then move to the next acupoint until all 6 acupoints were completed. The ear seed tapes were kept in place for 5 days and removed by participants for 2 days. After the 2-day rest period, the participant returned to the researcher to have the ear tapes replaced. Unilateral auricular points were used for the intervention and the treatment ear was changed to the other ear every week until the 3-week intervention was completed. All the auricular acupressure interventions were conducted by the same researcher.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a child (less than 18 years old) who was newly diagnosed with cancer (less than 3 months).
* parent of a child and who was receiving treatment with chemotherapy Must be able to swallow tablets

Exclusion Criteria:

* Parents were receiving any medication or treatment for insomnia.
* Parents had received any acupuncture or acupressure in the recent 3 months.
* Parents had ever been diagnosed with other chronic illnesses (such as cancer, heart disease, or asthma) at the time of data collection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Sleep Quality at baseline | Data were collected before auricular acupressure intervention
  The Pittsburgh Sleep Quality Index (PSQI) is a validated multidimensional measure that assesses individuals' sleep quality.
Sleep Quality at week 1 | Data were collected in the first week after completing 5 days of auricular acupressure.
  The Pittsburgh Sleep Quality Index (PSQI) is a validated multidimensional measure that assesses individuals' sleep quality.
Sleep Quality at week 2 | Data were collected in the second week after auricular acupressure interventtion.
  The Pittsburgh Sleep Quality Index (PSQI) is a validated multidimensional measure that assesses individuals' sleep quality.
Sleep Quality at week 3 | Data were collected in the 3rd week after auricular acupressure interventtion.
  The Pittsburgh Sleep Quality Index (PSQI) is a validated multidimensional measure that assesses individuals' sleep quality.

SECONDARY OUTCOMES:
Mood State at baseline | Data were collected before auricular acupressure intervention
  The Profile of Mood State (POMS) was developed to investigate individuals' mood status.
Mood State at week 1 | Data were collected in the first week after completing 5 days of auricular acupressure.
  The Profile of Mood State (POMS) was developed to investigate individuals' mood status.
Mood State at week 2 | Data were collected in the second week after auricular acupressure interventtion.
  The Profile of Mood State (POMS) was developed to investigate individuals' mood status.
Mood State at week 3 | Data were collected in the 3rd week after auricular acupressure interventtion.
  The Profile of Mood State (POMS) was developed to investigate individuals' mood status.
Quality of Life Short-Form at baseline | Data were collected before auricular acupressure intervention
  The Quality of Life Short-Form 36 (QOL-SF) was used to measure quality of life in parents of children with cancer for this study.
Quality of Life Short-Form at week 1 | Data were collected in the first week after completing 5 days of auricular acupressure.
  The Quality of Life Short-Form 36 (QOL-SF) was used to measure quality of life in parents of children with cancer for this study.
Quality of Life Short-Form at week 2 | Data were collected in the second week after auricular acupressure interventtion.
  The Quality of Life Short-Form 36 (QOL-SF) was used to measure quality of life in parents of children with cancer for this study.
Quality of Life Short-Form at week 3 | Data were collected in the 3rd week after auricular acupressure interventtion.
  The Quality of Life Short-Form 36 (QOL-SF) was used to measure quality of life in parents of children with cancer for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Chien Chiang, PhD, Principal Investigator — Chang Gung University of Science and Technology
Locations (1):
- Yi-Chien Chiang, Taoyuan District, Taoyuan City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chiang YC, Chen SH, Moser DK, Wen YC, Lin YT, Hsiao YC. Effectiveness of auricular acupressure in managing sleep quality, mood, and quality of life in parents of children with cancer: A pilot randomized controlled trial. Asia Pac J Oncol Nurs. 2024 Sep 25;11(11):100601. doi: 10.1016/j.apjon.2024.100601. eCollection 2024 Nov. PMID 39582551